CLINICAL TRIAL: NCT06856330
Title: Efficacy of Two Flap Palatoplasty (TFP) Versus Furlow With Buccinator Flap (FPBF) During Primary Palatoplasty on the Speech Development
Brief Title: Effect of Furlow Palatoplasty With Buccal Myomucosal Flap on the Speech Development
Status: Recruiting | Type: Observational
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Shaimaa Mohsen, associate professor of oral and maxillofacial surgery, Fayoum University
Other Study IDs: 55
Record Dates: First submitted 2025-02-22; First posted 2025-03-04 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Cleft Palate
MeSH Terms: conditions — Cleft Palate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- two flap palatoplasty group
  Interventions: Procedure: two flap palatoplasty
- furlow with buccal myomucosal flap group
  Interventions: Procedure: furlow with buccal myomucosal flap

INTERVENTIONS:
Procedure: furlow with buccal myomucosal flap — patients were treated with furlow with buccal myomucosal flap
  Groups: furlow with buccal myomucosal flap group
Procedure: two flap palatoplasty — patients were treated with two flap palatoplasty
  Groups: two flap palatoplasty group

SUMMARY:
About 20 patient will be collected according to the eligibility criteria and grouped into Group I : 10 patients were treated with furlow with buccinators flap Group II : 10 patients were treated with 2 flap palatoplasty All patients will be examined by an expert Phoniatrician by Recording of speech samples in Arabic language for the children in a soundproof room including repeated syllables, sentences with high-pressure sounds and counting from 1 to 10. The records will be analyzed to assess the degree of hypernasality, speech intelligibility and compensatory speech errors

ELIGIBILITY:
Inclusion Criteria:

* 3-5 years old childreen with previous treated complete cleft lip and palate, nonsyndromic.
* lip and palate repair performed by one craniofacial surgeon

Exclusion Criteria:

* Patients with syndromic cleft lip.
* Redu cases
* Bilateral cleft lip
* Patient older 5years or younger 3 years.
* Associated Cardiac anomalies.
* Any systemic condition

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 3-5 year old children with treated cleft palate
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-07-25 (Estimated)

PRIMARY OUTCOMES:
nasopharyngoscopic examination | through study completion, an average one week
  this will be done through the nasopharyngoscopic examination of the cleft patients after repair with Furlow with buccinator flap versus two flap palatoplasty. it will assess the grade of velopharyngeal closure during speech

CONTACTS AND LOCATIONS:
Locations (1):
- Fayoum University, Al Fayyum, Egypt

REFERENCES:
- [Derived] Refahee SM, Aboulhassan MA, Elrouby IM, Abd-El-Ghafour M. Speech outcome following primary furlow palatoplasty with buccal myomucosal flap versus two flap palatoplasty in patients with cleft palate. Clin Oral Investig. 2025 Dec 20;30(1):19. doi: 10.1007/s00784-025-06695-6. PMID 41420755